CLINICAL TRIAL: NCT01683071
Title: A Multicenter, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled, Dose Ranging Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of Single Injection Femoral Nerve Block With Liposome Bupivacaine for Postsurgical Analgesia in Subjects Undergoing Total Knee Arthroplasty
Brief Title: Femoral Nerve Block With Liposome Bupivacaine for Postsurgical Analgesia Following Total Knee Arthroplasty
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 402-C-323
Record Dates: First submitted 2012-09-07; First posted 2012-09-11 (Estimated); Results first posted 2020-12-09 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-11

CONDITIONS: Postoperative Pain
Keywords: Total knee arthroplasty; Analgesia; Pain management
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- (Part 1) EXPAREL 67 mg (Experimental): 5 mL EXPAREL (bupivacaine liposome injectable suspension) expanded with 15 mL normal saline as single-injection femoral nerve block ≤2 h preoperatively
  Interventions: Drug: EXPAREL 67 mg
- (Part 1) EXPAREL 133 mg (Experimental): 10 mL EXPAREL (bupivacaine liposome injectable suspension) expanded with 10 mL normal saline as single-injection femoral nerve block ≤2 h preoperatively
  Interventions: Drug: EXPAREL 133 mg
- (Part 1) EXPAREL 266 mg (Experimental): 20 mL EXPAREL (bupivacaine liposome injectable suspension) as single-injection femoral nerve block ≤2 h preoperatively
  Interventions: Drug: EXPAREL 266 mg
- (Part 1) Placebo (Placebo Comparator): 20 mL normal saline as single-injection femoral nerve block ≤2 h preoperatively
  Interventions: Drug: Placebo
- (Part 2) EXPAREL 266 mg (Experimental): 20 mL EXPAREL (bupivacaine liposome injectable suspension) as single-injection femoral nerve block ≤2 h preoperatively
  Interventions: Drug: EXPAREL 266 mg
- (Part 2) Placebo (Placebo Comparator): 20 mL normal saline as single-injection femoral nerve block ≤2 h preoperatively
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Normal saline 20 mL as single-injection femoral nerve block prior to total knee arthroplasty
  Other Names: Preservative-free normal saline.
  Arms: (Part 1) Placebo; (Part 2) Placebo
Drug: EXPAREL 67 mg — 5 mL EXPAREL expanded with 15 mL normal saline as single-injection femoral nerve block prior to total knee arthroplasty
  Other Names: Bupivacaine liposome injectable suspension 67 mg/5 mL
  Arms: (Part 1) EXPAREL 67 mg
Drug: EXPAREL 133 mg — 10 mL EXPAREL expanded with 10 mL normal saline as single-injection femoral nerve block prior to total knee arthroplasty
  Other Names: Bupivacaine liposome injectable suspension 133 mg/10 mL
  Arms: (Part 1) EXPAREL 133 mg
Drug: EXPAREL 266 mg — 20 mL EXPAREL as single-injection femoral nerve block prior to total knee arthroplasty
  Other Names: Bupivacaine liposome injectable suspension 266 mg/20 mL
  Arms: (Part 1) EXPAREL 266 mg; (Part 2) EXPAREL 266 mg

SUMMARY:
The primary objectives of Part 1 are to (1) evaluate three dose levels of liposome bupivacaine versus placebo with respect to the magnitude and duration of the analgesic effect achieved following single dose injection femoral nerve block with liposome bupivacaine, and (2) select a single therapeutic dose of liposome bupivacaine from the three dose levels to be tested in Part 2.

Part 2: The primary objective of Part 2 is to compare the magnitude and duration of the analgesic effect of single injection femoral nerve block of a single dose level of liposome bupivacaine (selected from Part 1) with placebo (preservative-free normal saline).

DETAILED DESCRIPTION:
This is a Phase 2/3, multicenter, randomized, double-blind, parallel-group, placebo-controlled, dose-ranging study in subjects undergoing primary unilateral total knee arthroplasty (TKA) under general or spinal anesthesia. Note: Bupivacaine cannot be used as the spinal anesthetic.

Part 1 During Part 1 of the study, approximately 100 subjects (25 per treatment arm) will be randomized to receive a single dose injection femoral nerve block with either one of three doses of liposome bupivacaine (67, 133, or 266 mg) or placebo in 20 mL under ultrasound guidance. Preservative-free normal saline will be added to the 67 mg and 133 mg doses of study drug to achieve a volume of 20 mL.

Part 2 In Part 2 of the study, approximately 180 subjects (randomized 1:1, resulting in approximately 90 liposome bupivacaine subjects and 90 placebo subjects) will receive a single dose injection femoral nerve block with the selected dose level of liposome bupivacaine (i.e., 67, 133, or 266 mg) or placebo in 20 mL under ultrasound guidance.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, >=18 years of age.
2. Scheduled to undergo primary unilateral TKA under general or spinal anesthesia.
3. American Society of Anesthesiologists (ASA) Physical Status 1, 2, or 3.
4. Able to demonstrate motor function by performing a 20-meter walk, unassisted with the optional use of a 4-legged walker, and sensory function by exhibiting sensitivity to cold.
5. Able to provide informed consent, adhere to the study visit schedule, and complete all study assessments.

Exclusion Criteria:

1. Currently pregnant, nursing, or planning to become pregnant during the study or within 1 month after study drug administration. Female subjects must be surgically sterile, at least 2 years menopausal, or using an acceptable method of birth control.

   If of childbearing potential, must have a documented negative pregnancy test within 24 hours before surgery.
2. Planned concurrent surgical procedure (e.g., bilateral TKA).
3. Use of any of the following medications within the times specified before surgery:

   long-acting opioid medication, NSAIDs, aspirin (except for low-dose aspirin used for cardioprotection) or acetaminophen within 3 days, or and any opioid medication within 24 hours.
4. Concurrent painful physical condition or concurrent surgery that may require analgesic treatment (such as an NSAID or opioid) in the postsurgical period for pain that is not strictly related to the surgical site administered study treatment, and which may confound the postsurgical assessments (e.g., significant pain from other joints including the non-index knee joint, chronic neuropathic pain, prior contralateral TKA, concurrent foot surgery).
5. Initiation of treatment with any of the following medications within 1 month of study drug administration or if the medication(s) are being given to control pain: selective serotonin reuptake inhibitors (SSRIs), selective norepinepherine reuptake inhibitors (SNRIs), gabapentin, pregabalin (Lyrica®), or duloxetine (Cymbalta®).
6. Current use of systemic glucocorticosteroids within 1 month of enrollment in this study.
7. Body weight < 50 kilograms (110 pounds) or a body mass index ≥ 40 kg/m2.
8. Contraindication to hydromorphone, oxycodone, or bupivacaine.
9. Administration of an investigational drug within 30 days or 5 elimination half-lives of such investigational drug, whichever is longer, prior to study drug administration, or planned administration of another investigational product or procedure during the subject's participation in this study.
10. Previous participation in a liposome bupivacaine study.
11. History of, suspected, or known addiction to or abuse of illicit drug(s), prescription medicine(s), or alcohol within the past 2 years.
12. Failure to pass the urine drug screen.
13. Uncontrolled anxiety, schizophrenia, or other psychiatric disorder that, in the opinion of the Investigator, could interfere with study assessments or compliance.
14. Malignancy in the last 2 years, with the exception of non-metastatic basal cell or squamous cell carcinoma of the skin or localized carcinoma in situ of the cervix.
15. Current or historical evidence of any clinically significant disease or condition, especially cardiovascular or neurological conditions that, in the opinion of the Investigator, may increase the risk of surgery or complicate the subject's postsurgical course.
16. Significant medical conditions or laboratory results that, in the opinion of the Investigator, indicate an increased vulnerability to study drugs and procedures.
17. Subjects who are planned to receive Entereg® (alvimopan).
18. Subjects who will receive prophylactic antiemetics or planned postsurgical antiemetics given without regard to the subject's emesis needs.
19. Use of dexmedetomidine HCl (Precedex®) within 3 days of surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 297 (Actual)
Dates: Start 2012-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erol Onel, MD, Study Director — Pacira Pharmaceuticals, Inc
Locations (30):
- United States (30):
  - ACHIEVE CLINICAL RESEARCH LLC 2017 Canyon Road Suite 41, Birmingham, Alabama
  - HORIZON RESEARCH GROUP INC 3610 Springhill Memorial Dr. N, Mobile, Alabama
  - Veritas Research, LLC, Mobile, Alabama
  - SHOALS MEDICAL TRIALS INC. 1300 S Montgomery Ave, Sheffield, Alabama
  - PHOENIX ORTHOPAEDIC SURGEONS 2525 W. Greenway Road Suite 114, Phoenix, Arizona
  - ALLIANCE RESEARCH CENTERS 24411 Health Center Drive Suite 350, Laguna Hills, California
  - ORTHOPADIC SURGERY Loma Linda University Health Care Dept. Pf Orthopaedic Surgery 250 East Caroline Street Suite A, San Bernardino, California
  - University of California, San Diego, San Diego, California
  - Ilfeld, Brian (Thornton) UNIVERSITY OF CALIFORNIA, SAN DIEGO 10610 Hunters Glen Drive, San Diego, California
  - FLORIDA RESEARCH ASSOCIATES, LLC / FLORIDA ORTHOPAEDIC ASSOCIATES 740 W. Plymouth Ave, DeLand, Florida
  - JACKSON MEMORIAL HOSPITAL UNVERSITY OF MIAMI 1611 Nw. 12th Ave C300, Miami, Florida
  - PENSACOLA RESEARCH CONSULTANTS,INC 5149 N.9th Avenue Suite 241, Pensacola, Florida
  - SHERIDAN CLINICAL RESEARCH, INC. 1613 N. Harrison Parkway Building C Suite 200, Sunrise, Florida
  - PHOENIX CLINICAL RESEARCH,LLC 7171 N. University Drive Suite 100, Tamarac, Florida
  - UNIVERSITY OF KANSAS HOSPITAL & MEDICAL CENTER Dept. Of Anesthesiology 3901 Rainbow Blvd. Ms 1034, Kansas City, Kansas
  - BEAUMONT HEALTH SYSTEM 44201 Dequindre Road Suite Pob 120, Troy, Michigan
  - COOPER UNIVERSITY HOSPITAL 1 Cooper Plaza 202 Dorrance Building, Camden, New Jersey
  - UNIVERSITY OF MEDICINE AND DENSITRY OF NEW JERSEY/NEW JERSEY MEDICAL SCHOOL 185 South Orange Ave. Department of Anesthesiology - MSB E538, Newark, New Jersey
  - NORTHERN WESTCHESTER HOSPTIAL Department Of Clinical Trials 400 East Main St., Mount Kisco, New York
  - ST. LUKE-ROOSEVELT HOSPITAL CENTER Dept. Of Anesthesiology 1111 Amsterdam Ave. Travis Bld. 7, New York, New York
  - INSALL-SCOTT-KELLY INSTITUTE 210 East 64th Street, New York, New York
  - UNIVERSITY OF NORTH CAROLINA AT CHAPEL HILL Department Of Anesthesiology 101 Manning Drive N0021, Cb 7010, Chapel Hill, North Carolina
  - CLEVELAND CLINIC FAIRVIEW HOSPTIAL 1801 Lorain Avenue, Cleveland, Ohio
  - CLEVELAND CLINIC 9500 Euclid Ave P-77, Cleveland, Ohio
  - PENN STATE MILTON S. HERSHEY MEDICAL CENTER H187,500 University Drive, Hershey, Pennsylvania
  - THOMAS JEFFERSON UNIVERSITY Dept. Of Anesthesiology 111 S. 11th Street Suite G 8490, Philadelphia, Pennsylvania
  - UPMC PRESBYTERIAN SHADYSIDE/ DEPT. OF ANESTHESIOLOGY POSNER PAIN CENTER 532 South Aiken Avenue Suite 407, Pittsburgh, Pennsylvania
  - UNIVERSITY OF TEXAS MEDICAL BRANCH Dept. Chairman, Orthopedic Surgery & Rehabilitation 2.316 Rebecca Sealy Hospital 301 University Blvd., Galveston, Texas
  - RESEARCH CONCEPTS,GP LLC 921 Gessner Rd. Anesthesia Dept., Classroom F, Houston, Texas
  - CHRISTUS ST. JOHN HOSPITAL 18300 St. John Dr., 2nd Floor, Surgery, Nassau Bay, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between September 24, 2012 and December 20, 2013 at 23 sites in the US
Pre-assignment Details: An unblinded dose selection committee reviewed Part 1 results for the primary endpoint, total postsurgical opioid consumption, time to first opioid rescue, and safety data, and recommended a dose level and sample size for Part 2.
Period: Part 1
Arm/Group | (Part 1) EXPAREL 67 mg | (Part 1) EXPAREL 133 mg | (Part 1) EXPAREL 266 mg | (Part 1) Placebo | (Part 2) EXPAREL 266 mg | (Part 2) Placebo
Started | 25 | 26 | 25 | 25 | 0 | 0
Completed | 21 | 22 | 22 | 20 | 0 | 0
Not Completed | 4 | 4 | 3 | 5 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 2 | 1 | 0 | 0
Not completed — Surgery Cancelled | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Did not receive study drug | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Early termination; met exclusion criteria | 0 | 2 | 1 | 0 | 0 | 0
Period: Part 2
Arm/Group | (Part 1) EXPAREL 67 mg | (Part 1) EXPAREL 133 mg | (Part 1) EXPAREL 266 mg | (Part 1) Placebo | (Part 2) EXPAREL 266 mg | (Part 2) Placebo
Started | 0 | 0 | 0 | 0 | 99 | 97
Completed | 0 | 0 | 0 | 0 | 82 | 82
Not Completed | 0 | 0 | 0 | 0 | 17 | 15
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 3 | 4
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 3 | 3
Not completed — Surgery cancelled | 0 | 0 | 0 | 0 | 4 | 2
Not completed — Did not receive study drug | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Met exclusion criterion | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Protocol deviation | 0 | 0 | 0 | 0 | 1 | 2
Not completed — Withdrawal by investigator decision | 0 | 0 | 0 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received study drug, with analysis by actual treatment received.
Groups:
- Total: Total of all reporting groups
Arm/Group | (Part 1) EXPAREL 67 mg | (Part 1) EXPAREL 133 mg | (Part 1) EXPAREL 266 mg | (Part 1) Placebo | (Part 2) EXPAREL 266 mg | (Part 2) Placebo | Total
Number analyzed (Participants) | 22 | 24 | 24 | 24 | 92 | 92 | 278
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.5 (8.41) | 65.7 (7.30) | 66.4 (8.94) | 66.1 (12.17) | 66.4 (10.35) | 63.6 (8.76) | 65.0 (9.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 16 | 14 | 14 | 52 | 57 | 161
  Male | 14 | 8 | 10 | 10 | 40 | 35 | 117
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2 | 3 | 8 | 9 | 24
  Not Hispanic or Latino | 21 | 23 | 22 | 21 | 84 | 83 | 254
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Asian | 1 | 0 | 1 | 0 | 2 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 2 | 4 | 15 | 14 | 38
  White | 20 | 22 | 21 | 20 | 75 | 76 | 234
  More than one race | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 22 | 24 | 24 | 24 | 92 | 92 | 278
American Society of Anesthesiologists (ASA) classification [Count of Participants; unit: Participants] — ASA classification: 1=normal healthy patient; 2=patient with mild systemic disease; 3=patient with severe systemic disease; 4=patient with severe systemic disease that is a constant threat to life; 5=a moribund patient who is not expected to survive without the operation; 6=a declared brain-dead patient whose organs are being removed for donor purposes.
  Participants
    1 | 0 | 0 | 1 | 0 | 7 | 3 | 11
    2 | 11 | 16 | 13 | 15 | 38 | 49 | 142
    3 | 11 | 8 | 10 | 9 | 47 | 40 | 125
    >/= 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Type of Anesthesia [Count of Participants; unit: Participants] — Population: One participant in the Part 2 placebo group did not have type of anesthesia recorded and therefore was not included in this analysis.
  Participants
    number analyzed (Participants) | 22 | 24 | 24 | 24 | 92 | 91 | 277
    General | 15 | 17 | 12 | 21 | 62 | 56 | 183
    Spinal | 6 | 7 | 12 | 3 | 28 | 35 | 91
    Other | 1 | 0 | 0 | 0 | 2 | 0 | 3
Duration of Surgery [Mean (Standard Deviation); unit: minutes] — Population: One participant in the Part 2 placebo group did not have duration of surgery recorded and therefore was not included in this analysis.
  minutes
    number analyzed (Participants) | 22 | 24 | 24 | 24 | 92 | 91 | 277
    (all) | 85.8 (25.53) | 88.5 (27.96) | 96.0 (37.94) | 85.0 (35.53) | 94.1 (34.43) | 94.9 (37.54) | 94.5 (35.9)
Incision length [Mean (Standard Deviation); unit: cm] — Population: One participant in the Part 1 EXPAREL 266 mg group, one participant in the Part 2 EXPAREL 266 mg group, and three participants in the Part 2 placebo group did not have incision length recorded and therefore were not included in this analysis.
  cm
    number analyzed (Participants) | 22 | 24 | 23 | 24 | 91 | 89 | 273
    (all) | 16.51 (2.457) | 14.98 (3.650) | 15.23 (2.834) | 18.25 (3.870) | 16.92 (4.987) | 16.29 (5.189) | 16.6 (5.08)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) of Numeric Rating Scale at Rest (NRS-R) Pain Intensity Scores Through 72 Hours
Description: AUC of NRS-R pain intensity scores through 72 hours. Pain intensity scores were measured on an 11-point NRS (0=no pain and 10=worst possible pain)
Time Frame: 0-72 hours
Population: Efficacy population: all participants in the safety analysis set who underwent the planned surgery, with analysis based on randomized treatment (regardless of treatment received)
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale * hr
Groups:
- (Part 1) EXPAREL 67 mg: 5 mL EXPAREL (bupivacaine liposome injectable suspension) expanded with 15 mL normal saline as single-injection femoral nerve block ≤2 h preoperatively
  EXPAREL: EXPAREL 67 mg, 133 mg, or 266 mg
- (Part 1) EXPAREL 133 mg: 10 mL EXPAREL (bupivacaine liposome injectable suspension) expanded with 10 mL normal saline as single-injection femoral nerve block ≤2 h preoperatively
  EXPAREL: EXPAREL 67 mg, 133 mg, or 266 mg
- (Part 1) EXPAREL 266 mg; (Part 2) EXPAREL 266 mg: 20 mL EXPAREL (bupivacaine liposome injectable suspension) as single-injection femoral nerve block ≤2 h preoperatively
  EXPAREL: EXPAREL 67 mg, 133 mg, or 266 mg
- (Part 1) Placebo; (Part 2) Placebo: 20 mL normal saline as single-injection femoral nerve block ≤2 h preoperatively
  Placebo: Normal saline 20 mL
Arm/Group | (Part 1) EXPAREL 67 mg | (Part 1) EXPAREL 133 mg | (Part 1) EXPAREL 266 mg | (Part 1) Placebo | (Part 2) EXPAREL 266 mg | (Part 2) Placebo
Number analyzed (Participants) | 22 | 24 | 24 | 24 | 92 | 91
score on a scale * hr | 533.4 (33.15) | 427.2 (31.73) | 436.2 (31.79) | 530.5 (31.73) | 418.9 (16.86) | 515.5 (16.95)
Statistical Analysis 1: Comparison: (Part 1) EXPAREL 67 mg vs (Part 1) Placebo; Test type: Superiority; p = 0.9494, ANCOVA; LSMD = 2.9, 95% CI 2-sided [-88 to 94]
Statistical Analysis 2: Comparison: (Part 1) EXPAREL 133 mg vs (Part 1) Placebo; Test type: Superiority; p = 0.0237, ANCOVA; LSMD = -103.3, 95% CI 2-sided [-192 to -14]
Statistical Analysis 3: Comparison: (Part 1) EXPAREL 266 mg vs (Part 1) Placebo; Test type: Superiority; p = 0.0386, ANCOVA; LSMD = -94.3, 95% CI 2-sided [-184 to -5]
Statistical Analysis 4: Comparison: (Part 2) EXPAREL 266 mg vs (Part 2) Placebo; Test type: Superiority; p < 0.0001, ANCOVA; LSMD = -96.5, 95% CI 2-sided [-144 to -49]

2. Secondary Outcome: Total Postsurgical Opioid Consumption Through 72 Hours
Description: Total postsurgical opioid consumption of opioid rescue pain medication (converted to IV morphine equivalents) through 72 hours
Time Frame: 0-72 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg morphine equivalents
Arm/Group | (Part 1) EXPAREL 67 mg | (Part 1) EXPAREL 133 mg | (Part 1) EXPAREL 266 mg | (Part 1) Placebo | (Part 2) EXPAREL 266 mg | (Part 2) Placebo
Number analyzed (Participants) | 22 | 24 | 24 | 24 | 92 | 91
mg morphine equivalents | 126.69 (75.972) | 100.35 (53.177) | 105.96 (53.402) | 124.78 (58.743) | 93.19 (58.133) | 122.08 (70.312)
Statistical Analysis 1: Comparison: (Part 1) EXPAREL 67 mg vs (Part 1) Placebo; Test type: Superiority; p = 0.6182, ANOVA; Geometric LSM ratio = 0.90, 95% CI 2-sided [0.6 to 1.3]
Statistical Analysis 2: Comparison: (Part 1) EXPAREL 133 mg vs (Part 1) Placebo; Test type: Superiority; p = 0.1097, ANOVA; Geometric LSM ratio = 0.73, 95% CI 2-sided [0.5 to 1.1]
Statistical Analysis 3: Comparison: (Part 1) EXPAREL 266 mg vs (Part 1) Placebo; Test type: Superiority; p = 0.4046, ANOVA; Geometric LSM ratio = 0.85, 95% CI 2-sided [0.6 to 1.3]
Statistical Analysis 4: Comparison: (Part 2) EXPAREL 266 mg vs (Part 2) Placebo; Test type: Superiority; p = 0.0016, ANOVA; Geometric LSM ratio = 0.74, 95% CI 2-sided [0.6 to 0.9]

3. Secondary Outcome: Time to First Opioid Rescue Through 72 Hours
Description: Time to first opioid rescue medication consumed through 72 hours
Time Frame: 0-72 hours
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | (Part 1) EXPAREL 67 mg | (Part 1) EXPAREL 133 mg | (Part 1) EXPAREL 266 mg | (Part 1) Placebo | (Part 2) EXPAREL 266 mg | (Part 2) Placebo
Number analyzed (Participants) | 22 | 24 | 24 | 24 | 92 | 91
hours | 0.49 [0.300 to 0.650] | 0.37 [0.283 to 0.700] | 1.29 [0.367 to 2.350] | 0.41 [0.300 to 0.550] | 0.44 [0.400 to 0.533] | 0.43 [0.367 to 0.567]

ADVERSE EVENTS:
Time Frame: From screening through postsurgical day 30
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans whether or not considered drug-related. An AE could therefore have been any unfavorable and unintended sign (eg, abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug without any judgment about causality.
  Serious AEs were defined as per clinicaltrials.gov.
  The safety analysis set includes all subjects who received study drug, based on treatment received.
Arm/Group | (Part 1) EXPAREL 67 mg | (Part 1) EXPAREL 133 mg | (Part 1) EXPAREL 266 mg | (Part 1) Placebo | (Part 2) EXPAREL 266 mg | (Part 2) Placebo
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/24 | 0/24 | 0/24 | 0/92 | 0/92
Serious Adverse Events (participants affected / at risk) | 4/22 | 2/24 | 1/24 | 3/24 | 8/92 | 9/92
Other Adverse Events (participants affected / at risk) | 19/22 | 20/24 | 21/24 | 21/24 | 82/92 | 83/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | (Part 1) EXPAREL 67 mg (N=22) | (Part 1) EXPAREL 133 mg (N=24) | (Part 1) EXPAREL 266 mg (N=24) | (Part 1) Placebo (N=24) | (Part 2) EXPAREL 266 mg (N=92) | (Part 2) Placebo (N=92)
Anemia (Blood and lymphatic system disorders) | 2 | 0 | 1 | 0 | 1 | 2
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Device Related Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Wound Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Wound Dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0
Wound Decomposition (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Wound Necrosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Local Swelling (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Acute Prerenal Failure (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 4 | 1
Edema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Systemic Inflammatory Response Syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypovolemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Orthostatic Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1
Cardiac Failure Congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Type IV Hypersensitivity Reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | (Part 1) EXPAREL 67 mg (N=22) | (Part 1) EXPAREL 133 mg (N=24) | (Part 1) EXPAREL 266 mg (N=24) | (Part 1) Placebo (N=24) | (Part 2) EXPAREL 266 mg (N=92) | (Part 2) Placebo (N=92)
Nausea (Gastrointestinal disorders) | 8 | 14 | 13 | 9 | 49 | 61
Constipation (Gastrointestinal disorders) | 3 | 2 | 6 | 1 | 32 | 32
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 2 | 26 | 38
Pyrexia (General disorders) | 8 | 7 | 8 | 3 | 28 | 24
Dizziness (Nervous system disorders) | 3 | 3 | 4 | 6 | 15 | 19
Headache (Nervous system disorders) | 1 | 3 | 2 | 1 | 5 | 4
Tremor (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 4 | 1 | 4 | 2 | 8 | 5
Insomnia (Psychiatric disorders) | 1 | 2 | 2 | 4 | 5 | 11
Confusional State (Psychiatric disorders) | 1 | 2 | 0 | 0 | 3 | 3
Pruritis (Skin and subcutaneous tissue disorders) | 1 | 2 | 2 | 2 | 33 | 31
Pruritis Generalized (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 3 | 2 | 2
Procedural Hypotension (Injury, poisoning and procedural complications) | 2 | 2 | 3 | 0 | 10 | 6
Wound Dehiscence (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 1 | 2 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 2 | 3 | 6
Hypotension (Vascular disorders) | 1 | 2 | 0 | 0 | 3 | 8
Cellulitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 1
Body Temperature Increased (Investigations) | 0 | 0 | 2 | 0 | 6 | 4
Feeling Cold (General disorders) | 0 | 0 | 1 | 0 | 9 | 8
Local Swelling (General disorders) | 0 | 1 | 0 | 0 | 6 | 5
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 10 | 11
Anemia Postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 6 | 9
Urinary Retention (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 12 | 6
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 5 | 6
Mobility Decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 6 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results conducted at Site shall not be published before 1st multicenter publication by Sponsor but can proceed if there is no such publication ≤18 months after study completion/termination at all sites and all data have been received. Before submitting manuscript/materials to an outside person/entity, site shall give Sponsor 60 days to review and comment. Site shall, upon request, further delay publication/presentation for ≤120 days to allow Sponsor to protect its interests in Inventions.

DOCUMENTS (2):
  • Study Protocol (2013-04-19): https://cdn.clinicaltrials.gov/large-docs/71/NCT01683071/Prot_000.pdf
  • Statistical Analysis Plan (2013-12-09): https://cdn.clinicaltrials.gov/large-docs/71/NCT01683071/SAP_001.pdf